CLINICAL TRIAL: NCT05205980
Title: Motor Learning of Fall Resistant Skills From Laboratory-induced Falling Among People With Mild Alzheimer's Disease
Brief Title: Perturbation Training Reduces Falls in People With Alzheimer's Disease (AD)
Acronym: STAD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Georgia State University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Alzheimer's Association (Other)
Responsible Party: Principal Investigator, Feng Yang, PhD, Associate Professor, Georgia State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: H22487
Record Dates: First submitted 2021-12-15; First posted 2022-01-25 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The assessor will be blinded to the group assignment of each participant.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training group (Experimental): This arm will receive a single-session perturbation training treatment on a treadmill under the protection of a safety harness.
  Interventions: Behavioral: Perturbation training
- Control group (Sham Comparator): This arm will not receive perturbation training but will go through harnessed walking on the same treadmill for the same time as the other group.
  Interventions: Behavioral: Perturbation training

INTERVENTIONS:
Behavioral: Perturbation training — Participants will experience repeated perturbations mixed with non-perturbed trials on the treadmill with the protection by a harness.

SUMMARY:
This study will examine the overall capacity of people with Alzheimer's disease learning fall-resistant skills from perturbation training.

DETAILED DESCRIPTION:
Falls can cause injury and death in older adults. Those with Alzheimer's disease are at an even higher fall risk. Our goal is to test if people with mild Alzheimer's disease can learn fall prevention skills from the exposure to large-scale perturbations on a treadmill. Two groups with mild Alzheimer's disease will be enrolled. One group will attend a perturbation training session while the other group receives no training. Groups will then be exposed to perturbations on the ground immediately and three or six months after the training. Over six months after the training, daily-living falls will be tracked for both groups. The falls following the perturbations in the lab and daily-living all-cause falls will be compared between groups to test our specific aims: 1) to test if people with Alzheimer's disease can adapt to large-scale external perturbations and learn fall resistant motor skills; 2) to inspect whether people with Alzheimer's disease can retain motor skills learned in Aim 1; and 3) to determine if people with Alzheimer's disease can generalize fall resistant skills to different contexts (treadmill to overground, inside the lab to outside the lab).

ELIGIBILITY:
Inclusion Criteria:

* Participants must be at least 65 years old;
* Participants have a clinical diagnosis of probable AD;
* Participants can read and understand English;
* Participants must be able to walk independently at least 25 feet;
* Participants must be able to stand independently for at least 30 seconds;
* Participants must have a Montreal Cognitive Assessment score of 11-21 or Mini Mental Status Examination score between 18 and 23.

Exclusion Criteria:

* Individuals have ever experienced perturbation training;
* Individuals have hypotension or uncontrolled hypertension;
* Individuals exhibit osteoporosis;
* Participants suffer from coexisting psychiatric disorders, or other neurological conditions, or injuries, etc.

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-04-28 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Lab-induced faller rate | 6 months
  The outcome of each perturbation trial will be determined as a fall if the peak load cell force exceeds 30% of the body weight. The load cell records the force applied to the human body by the safety harness system after a perturbation. The lab-induced faller rate will be calculated as the ratio of the number of fallers to the number of participants within each group.

SECONDARY OUTCOMES:
Dynamic stability | 6 months
  Dynamic stability will be calculated for each perturbation trial based on the kinematics of the body's center of mass relative to the base of support.
Number of prospective fall incident | 6 months
  The number of all cause falls in daily-living activities after the training session will be recorded for each participant.

OTHER OUTCOMES:
Berg Balance Scale | 6 months
  Berg balance scale will be used to objectively determine a participant' ability (or inability) to safely balance during a series of preset tasks. The score of the Berg Balance Scale is between 0 and 56 with a higher value indicating a better balance ability.
Mobility | 6 months
  Functional mobility will be assessed using the Timed-Up-and-Go test. The time used to complete the test will be recorded. The shorter the time, the better mobility.
Muscle strength | 6 months
  Strength capacity will be tested on the knee joint as the maximum strength the knee joint can produce. The measurement will be taken on an isokinetic dynamometer.
Pressure sensation level | 6 months
  The tactile sensation level at the dominant sole will be determined as the number of sites where the participant can feel the pressure produced by the monofilament.
Posturography test | 6 months
  This test will be done when the participant is standing on a pair of force plates. The center of pressure movement will be calculated from the ground reaction force measured by the force plates. The center of pressure excursion in the anteroposterior and mediolateral directions will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Feng Yang, PhD, Principal Investigator — Georgia State University
Locations (1):
- Reminiscent, Valdosta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No